CLINICAL TRIAL: NCT06771726
Title: Multicenter Study Protocol: Research on Evaluation and Detec-tion of Surgical Wound Complications with AI-based Recogni-tion. (REDSCAR-trial)
Brief Title: Multicenter Study Protocol: Research on Evaluation and Detection of Surgical Wound Complications with AI-based Recognition. (REDSCAR-trial)
Acronym: REDSCAR
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitat de les Illes Balears (Other)
Responsible Party: Principal Investigator, Andrea Craus, Principal Investigator, Universitat de les Illes Balears
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IB 5087/22 PI; PID2020-113870GB-I00 (Other Grant/Funding Number: MCIN/AEI/10.13039/501100011033)
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Surgical Wound Infection
Keywords: surgical wound infection; Telemedicine; smartphone application; artificial intelligence
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: This multicenter prospective study uses a paired cohort design with a non-randomized, single-blinded approach, where each participant served as their own control. The investigators remain unaware of the application's recommendations dur-ing wound assessments. The study will include adult patients undergoing abdominal surgery at different hospitals. This study involves the use of the RedScar© app on pa-tients' smartphones. Patients will complete a brief health questionnaire and upload a wound photograph to the app, which will provide recommendations based on the risk of infection detected. Simultaneously, an in-person wound assessment will be con-ducted by the investigator to compare results.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Redscar app (Experimental): Telematic follow-up with App
  Interventions: Device: RedScar App
- In-Person (No Intervention): In-person visit to the clinics

INTERVENTIONS:
Device: RedScar App — use of the RedScar© app on patients' smartphones. Patients will complete a brief health questionnaire and upload a wound photograph to the app, which will provide recommendations based on the risk of infection detected. Simultaneously, an in-person wound assessment will be conducted by the investigator to compare results.
  Arms: Redscar app

SUMMARY:
The increasing use of telemedicine in surgical care has demonstrated significant poten-tial for improving patient outcomes and optimizing healthcare resources. This study investigates the efficacy of the RedScar© app in telematic detection and monitoring of surgical site infections (SSIs), a major cause of healthcare-associated infections (HAIs) with significant economic and health impacts. RedScar© leverages a patient's smartphone to provide automated infection risk assessments without requiring clini-cian input, offering a potential solution for remote postoperative care. In a pilot study, RedScar© demonstrated 100% sensitivity and 83.13% specificity in detecting SSIs, with high patient satisfaction regarding its comfort, cost-effectiveness, and ability to reduce absenteeism. This multicenter prospective study aims to validate these findings, com-paring app-based detection with in-person evaluations. Primary objectives include as-sessing the sensitivity and specificity of RedScar© using receiver operating character-istic (ROC) analysis, while secondary objectives include evaluating patient satisfaction and standardizing telematic follow-up across centers. The study will include 168 pa-tients undergoing abdominal surgery, with follow-up assessments conducted remotely via the app and in-person at specified intervals. Data will be analysed using descrip-tive and statistical methods to assess diagnostic accuracy and patient satisfaction. This research seeks to further develop RedScar© as a reliable, scalable tool for enhancing postoperative care, reducing healthcare costs, and improving patient experiences in surgical recovery.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have signed an informed consent.
* Participants must be over 18 years of age.
* Participants must have undergone either urgent or scheduled surgery performed via laparotomy or laparoscopy.
* Participants need access to a smartphone capable of downloading the app with android OS.
* Either the participant or a close family member must be able to operate the app effectively.
* Participants must be able to attend follow-up consultations at the surgical outpatient clinic after discharge, one week post-surgery, or earlier if the app flags a potential infection.

Exclusion Criteria:

* Patients who lack access to a smartphone or are unable to properly use the app.
* Patients unfamiliar with mobile devices or unable to comprehend the app's functionality or questions.
* Patients who did not provide informed consent.
* Patients who are unable to comply with the follow-up requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of RedScar App | "From enrollment to the end of treatment at 8 weeks"
  To assess the sensitivity and specificity of the RedScar© application for detecting wound infection, comparing the app with in-person diagnosis. The ROC curve will be used to analyze the overall performance of the app and identify the optimal cut-off for the "Red Proportion" (maximizing sensitivity and specificity).

SECONDARY OUTCOMES:
Satisfaction Asessment | From enrollment to the end of treatment at 8 weeks
  Assess the satisfaction level of subjects undergoing telemedicine-based follow-up using a validated telemedicine satisfaction questionnaire (Yip et al.). Minimum: 0. Maximum: 14. Higher scores mean a better satisfaction.

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital de Fuenlabrada, Madrid
  - Hospital Universitario Severo Ochoa, Madrid
  - Hospital General Mateu Orfila, Maó
  - Hospital Universitario Son Espases, Palma
  - Universidad Islas Baleares, Palma

IPD SHARING:
Plan to Share IPD: Yes
A virtual repository of surgical wound photographs was created and made available to other researchers. This repository can be accessed through the website redscar.uib.es
Supporting Information: Analytic Code
Time Frame: 2023-No limit
Access Criteria: Authorization must be granted via email.
URL: http://redscar.uib.es

REFERENCES:
- [Background] Craus-Miguel A, Munar M, Moya-Alcover G, Contreras-Nogales AM, Gonzalez-Hidalgo M, Segura-Sampedro JJ. Enhancing Surgical Wound Monitoring: A Paired Cohort Study Evaluating a New AI-Based Application for Automatic Detection of Potential Infections. J Clin Med. 2024 Dec 23;13(24):7863. doi: 10.3390/jcm13247863. PMID 39768786
- [Background] Segura-Sampedro JJ, Rivero-Belenchon I, Pino-Diaz V, Rodriguez Sanchez MC, Pareja-Ciuro F, Padillo-Ruiz J, Jimenez-Rodriguez RM. Feasibility and safety of surgical wound remote follow-up by smart phone in appendectomy: A pilot study. Ann Med Surg (Lond). 2017 Jul 18;21:58-62. doi: 10.1016/j.amsu.2017.07.040. eCollection 2017 Sep. PMID 28794868
- See also: RedScar Image Repository — http://redscar.uib.es/